CLINICAL TRIAL: NCT06734611
Title: Effectiveness Study of Folic Acid Fortified Iodized Salt to Increase Folate Concentrations in Women of Reproductive Age in Zambia, a Non-fortifying Country
Brief Title: Folic Acid Salt Study (FISFA Zambia)
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Collaborators: Centre for Infectious Disease Research in Zambia (Other); Baylor College of Medicine (Other)
Responsible Party: Principal Investigator, Anastasia Smith, Clinical Research Manager, University of Alabama at Birmingham
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: IRB-300013997; FISFA-Zambia-2025 (Other: University of Alabama at Birmingham)
Record Dates: First submitted 2024-12-10; First posted 2024-12-16 (Actual); Last update posted 2025-12-29 (Actual); Status verified 2025-12

CONDITIONS: Folate Deficiency; Neural Tube Defects
Keywords: folic acid; iodine; salt; serum folate; red blood cell folate; prevention; folate insufficiency; Malnutrition; Nervous System Malformations; Spinal Dysraphism; Vitamin B9; Micronutrients
MeSH Terms: conditions — Folic Acid Deficiency; Neural Tube Defects; Malnutrition; Nervous System Malformations; Spinal Dysraphism | interventions — Folic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- FISFA arm (Experimental): Dietary Supplement: fortified iodized salt with folic acid (FISFA)
  Interventions: Dietary Supplement: Fortified Iodized Salt with Folic Acid (FISFA)

INTERVENTIONS:
Dietary Supplement: Fortified Iodized Salt with Folic Acid (FISFA) — Addition of folic acid to iodized salt for daily consumption to assess folate levels.

SUMMARY:
Question: How effective is fortified iodized salt with folic acid (FISFA) in increasing serum and red blood cell folate in non-lactating, non-pregnant women of reproductive age in the country of Zambia who do not have active food fortification with a folic acid program?

Participants will:

* Consume salt with folic acid instead of their regular salt for 6 months
* Have a blood draw 4 times
* Fill out surveys

DETAILED DESCRIPTION:
The objective of this nonrandomized controlled intervention trial is to measure the effectiveness of fortified iodized salt with folic acid (FISFA) on increasing blood folate concentrations as a preventive measure against folate-sensitive neural tube defects (NTDs) in a non-fortifying country of Zambia.

The main questions it aims to answer are:

Aim 1: Measure the effectiveness of FISFA on increasing serum and red blood cell folate concentrations in women of reproductive age in a non-fortifying country.

Aim 2: Assess the risk of neural tube defects by measuring folate insufficiency levels via serum and red blood cell concentrations in women of reproductive age in a non-fortifying country.

Aim 3: Assess taste and color acceptability of FISFA by study population.

ELIGIBILITY:
Inclusion Criteria:

* Voluntary participation in the study
* Do not intend to get pregnant
* Not lactating or pregnant
* Live alone or with a partner if they can be compliant and not share the study salt.
* Aged between 18 and 45 years

Exclusion Criteria:

* Pregnant or lactating

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 250 (Estimated)
Dates: Start 2026-03-01 (Estimated); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Measure change in median and mean serum folate levels between baseline, month 1, month 3 and month 6 (endpoint) | 0-6 months
  Evaluate folate blood levels pre and post intervention
Measure change in median and mean red blood cell folate levels between baseline, month 1, month 3 and month 6 (endpoint) | 0-6 months
  Evaluate folate blood levels pre and post intervention

SECONDARY OUTCOMES:
Descriptive analysis of acceptability of FISFA by participants (taste and color on Likert scale) | 1,3,6 months
  Evaluate salt with folic acid acceptability using Likert scale (1-5, with 5 being the better outcome)
Measure of folate insufficiency via serum and RBC concentration | 0-6 months
  Comparing folate insufficiency via serum and RBC concentration to recommended levels of 25.5 nmol/L (serum) and 906 nmol/L in RBC for WRA

CONTACTS AND LOCATIONS:
Overall Officials: Anastasia A Smith, DrPH, Principal Investigator — University of Alabama at Birmingham
Locations (2):
- University of Alabama at Birmingham, Birmingham, Alabama, United States
- Centre for Infectious Disease Research in Zambia, Lusaka, Zambia

IPD SHARING:
Plan to Share IPD: No
Redacted information will be made available upon request.